CLINICAL TRIAL: NCT04695106
Title: Dual Antithrombotic Therapy With Dabigatran and Ticagrelor in Patients With Acute Coronary Syndrome and Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention (ADONIS-PCI)
Brief Title: Dual Antithrombotic Therapy With Dabigatran and Ticagrelor in Patients With ACS and Non-valvular AF Undergoing PCI
Acronym: ADONIS-PCI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Collaborators: Medical University of Warsaw (Other); Nicolaus Copernicus University (Other); National Institute of Cardiology, Warsaw, Poland (Other); Military Institute od Medicine National Research Institute (Other); Bielanski Hospital (Other); Medical University of Silesia (Other); Poznan University of Medical Sciences (Other); University of Opole, Poland (Unknown); Medical University of Łódź (Other); Voivodeship Hospital, Kielce, Poland (Unknown); Voivode Specialist Hospital in Olsztyn, Poland (Unknown); Medical University of Lublin (Other); Pomeranian Medical University Szczecin (Other); Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Milosz Jaguszewski MD PhD FESC, Professor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBK 182/1/2020; 2020-004887-24 (EudraCT Number)
Record Dates: First submitted 2020-11-25; First posted 2021-01-05 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation; Antithrombotic Therapy; Acute Coronary Syndrome; Percutaneous Coronary Interventions
Keywords: Atrial Fibrillation; Acute Coronary Syndrome; Dabigatran; Ticagrelor; Antithrombotic therapy
MeSH Terms: conditions — Atrial Fibrillation; Acute Coronary Syndrome | interventions — Ticagrelor; Dabigatran; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study population (Experimental): In the study group (both STEMI and NSTE-ACS), aspirin will be discontinued, and ticagrelor will be started at a loading dose of 180 mg, irrespective of timing and dosing of clopidogrel, and continued at a maintenance dose of 90 mg twice daily for 1 month, followed by 60 mg twice daily up to 12 months.
  Dabigatran will be used as a standard-of-care. Lower dose dabigatran (110 mg twice daily) will be used in patients ≥80 years of age and will be considered in patients (i) 75-80 years of age, (ii) with creatinine clearance 30-50 ml/min, (iii) at high risk of bleeding (HAS-BLED ≥ 3), (iv) at high-risk of gastrointestinal bleeding (with esophagitis, gastritis, gastroesophageal reflux disease), and (v) treated with verapamil, in accordance with the guidelines.
  Interventions: Drug: Ticagrelor; Drug: Dabigatran Etexilate
- Control group (Active Comparator): In the control group, aspirin and clopidogrel will be continued depending on the diagnosis (STEMI or NSTE-ACS) and bleeding risk. In patients with STEMI, aspirin will be discontinued after 1-6 months, according to a balance between the estimated risk of recurrent coronary events and bleeding. In patients at high bleeding risk aspirin will be discontinued after 1 month. Subsequently, all patients will be treated with clopidogrel and dabigatran up to 12 months. In the NSTE-ACS group, aspirin will be used up to 1 week (in-hospital period), extendable up to one month in patients at high ischaemic risk. Dual therapy will be continued up to 12 months with the possibility of shortening for patients at high bleeding risk.
  Dabigatran will be used as a standard-of-care (as above).
  Interventions: Drug: Dabigatran Etexilate; Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Within 72 hours post PCI, patients will be randomized in a 1:1 ratio to receive one of the two treatments: dual therapy with ticagrelor (90 mg twice daily for one month, followed by 60 mg twice daily up to 12 months) plus dabigatran (150 mg twice daily or 110 mg twice daily; standard of care) or triple therapy with clopidogrel (75 mg once daily) plus aspirin (75 mg once daily) plus dabigatran (150 mg twice daily or 110 mg twice daily), according to current guidelines. Study treatment will be continued for 12 months.
  Other Names: Brilique
  Arms: Study population
Drug: Dabigatran Etexilate — Within 72 hours post PCI, patients will be randomized in a 1:1 ratio to receive one of the two treatments: dual therapy with ticagrelor (90 mg twice daily for one month, followed by 60 mg twice daily up to 12 months) plus dabigatran (150 mg twice daily or 110 mg twice daily; standard of care) or triple therapy with clopidogrel (75 mg once daily) plus aspirin (75 mg once daily) plus dabigatran (150 mg twice daily or 110 mg twice daily), according to current guidelines. Study treatment will be continued for 12 months
  Other Names: Pradaxa
Drug: Aspirin — Within 72 hours post PCI, patients will be randomized in a 1:1 ratio to receive one of the two treatments: dual therapy with ticagrelor (90 mg twice daily for one month, followed by 60 mg twice daily up to 12 months) plus dabigatran (150 mg twice daily or 110 mg twice daily; standard of care) or triple therapy with clopidogrel (75 mg once daily) plus aspirin (75 mg once daily) plus dabigatran (150 mg twice daily or 110 mg twice daily), according to current guidelines. Study treatment will be continued for 12 months
  Arms: Control group
Drug: Clopidogrel — Within 72 hours post PCI, patients will be randomized in a 1:1 ratio to receive one of the two treatments: dual therapy with ticagrelor (90 mg twice daily for one month, followed by 60 mg twice daily up to 12 months) plus dabigatran (150 mg twice daily or 110 mg twice daily; standard of care) or triple therapy with clopidogrel (75 mg once daily) plus aspirin (75 mg once daily) plus dabigatran (150 mg twice daily or 110 mg twice daily), according to current guidelines. Study treatment will be continued for 12 months
  Arms: Control group

SUMMARY:
More than 25% of patients referred for diagnostic coronary angiography and percutaneous coronary intervention (PCI) due to acute coronary syndrome (ACS) suffer from non-valvular atrial fibrillation (AF). In this particular setting, balancing between the prevention of thrombosis and the risk of bleeding remains challenging. Oral anticoagulation (OAC) prevents stroke and systemic embolism, but has not been shown to prevent stent thrombosis (ST). Dual antiplatelet therapy (DAPT) reduces the incidence of recurrent ischemic events and ST, but is less effective in reducing the incidence of cardioembolic stroke associated with AF. A common guideline-supported practice is to combine three drugs (OAC, aspirin and clopidogrel) in a triple therapy, which is associated with high annual risk (up to 25%) of major bleeding. Thus, new therapeutic strategies are urgently needed to maintain the efficacy while improving the safety of treatment in patients with AF and ACS undergoing PCI.

This is a prospective, randomized, open-label, blinded-endpoint, non-inferiority trial. 2230 patients with non-valvular AF that had undergone successful PCI due to an ACS within the previous 72 hours will be randomized in 1:1 ratio to receive one of the two treatments: dual therapy with dabigatran (150 mg twice daily or 110 mg twice daily) and ticagrelor (90 mg twice daily for 1 month, followed by 60 mg twice daily up to 12 months), or standard therapy according to current guidelines triple therapy with dabigatran (150 mg b.i.d. or 110 mg b.i.d.) plus clopidogrel (75 mg o.d.) plus aspirin (75 mg o.d.) followed by double therapy depending on the bleeding and ischaemic risk. Study treatment will be continued for 12 months. The primary study end-point is the first major or clinically relevant non-major bleeding event (per ISTH), in a time-to-event analysis. The main secondary end-point is a composite efficacy end-point of thromboembolic events (myocardial infarction, stroke, or systemic embolism), death, or unplanned revascularization (PCI or coronary artery bypass grafting) at 12 months.

We expect that dual antithrombotic therapy including reduced dose ticagrelor and dabigatran is at least non-inferior regarding bleeding risk and ischaemic protection, compared to the standard triple therapy in patients with AF and after ACS, treated with PCI.

DETAILED DESCRIPTION:
Health problem More than 25% of patients referred for diagnostic coronary angiography and percutaneous coronary intervention (PCI) due to acute coronary syndrome (ACS) suffer from non-valvular atrial fibrillation (AF). In this particular setting, balancing between the prevention of thrombosis and the risk of bleeding remains challenging. Oral anticoagulation (OAC) prevents stroke and systemic embolism but does not prevent stent thrombosis. Dual antiplatelet therapy (DAPT) reduces the incidence of recurrent ischemic events and stent thrombosis but is less effective in reducing the incidence of cardioembolic stroke associated with AF. A common guideline-supported practice is to combine all three drugs (OAC, aspirin, and clopidogrel) in triple therapy, but this approach remains an expert opinion. Moreover, triple therapy is associated with a high annual risk (up to 25%) of major bleeding. Thus, new therapeutic strategies are urgently needed to maintain efficacy while improving treatment safety in patients with AF and ACS undergoing PCI. The investigators hypothesize that dual antithrombotic therapy, including reduced dose ticagrelor (study group, n=1115), is non-inferior regarding bleeding risk and ischaemic protection to the standard triple therapy (control group, n=1115) in patients with AF and treated with PCI due to ACS.

Study population The study's target population is male and female patients aged ≥18 years with non-valvular AF that underwent a successful PCI due to an ACS. AF may be paroxysmal, persistent or permanent but must not be secondary to a reversible disorder such as myocardial infarction, pulmonary embolism, recent surgery, pericarditis, or thyrotoxicosis. ACS may be ST-elevation myocardial infarction (STEMI), non-STEMI (NSTEMI), or unstable angina (UA).

Study design This is a multicentre, prospective, randomized, open-label, blinded endpoint, non-inferiority trial. Within 72 hours post PCI, patients will be randomized in a 1:1 ratio to receive one of the two treatments: dual therapy with ticagrelor (90 mg twice daily for one month, followed by 60 mg twice daily up to 12 months) plus dabigatran (150 mg twice daily or 110 mg twice daily; standard of care) or triple therapy with clopidogrel (75 mg once daily) plus aspirin (75 mg once daily) plus dabigatran (150 mg twice daily or 110 mg twice daily), according to current guidelines. Study treatment will be continued for 12 months.

Endpoints The primary study endpoint is the first major or clinically relevant non-major bleeding event, as defined by the International Society on Thrombosis and Haemostasis (ISTH), in a time-to-event analysis. The main secondary endpoint is a composite efficacy endpoint of thromboembolic events (myocardial infarction, stroke, or systemic embolism), death, or unplanned revascularization (PCI or coronary artery bypass grafting).

Expected results The investigators expect that the off-label regimen of dual antithrombotic therapy, including reduced dose ticagrelor, is at least non-inferior regarding bleeding risk and ischaemic protection, to the standard triple therapy in patients with AF and after ACS, treated with PCI.

Discussion The investigators propose a new off-label treatment regimen which is reduced dose ticagrelor in patients with AF and ACS. The most scientifically valuable points of the proposed project are the first-ever (i) attempt to administer the off-label potent P2Y12 inhibitor (ticagrelor) as a part of dual antiplatelet therapy in patients with AF and ACS and (ii) evaluation of the reduced dose of ticagrelor in the setting of ACS. The three most innovative aspects are: (i) new treatment regimen with a reduced ticagrelor dose in ACS setting, (ii) possibility to introduce the polypill containing ticagrelor and dabigatran to the Polish market, and (iii) potential manufacture of the polypill containing various doses of ticagrelor and dabigatran, depending on the patient's individual ischaemic and bleeding risk. If successful, the proposed study will answer the burning clinical question about the optimal treatment strategy in patients with AF and ACS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥18 years'
* Patients with new-onset or pre-existing non-valvular AF that have been receiving oral anticoagulant treatment with dabigatran for at least 48 hours or were treatment naïve prior to PCI. AF may be paroxysmal, persistent or permanent, but must not be secondary to a reversible disorder such as MI, pulmonary embolism, recent surgery, pericarditis or thyrotoxicosis unless long-term treatment with an OAC is anticipated.
* Patients presenting with ACS that had undergone a successful PCI with drug-eluting stent (DES) implantation within the previous 72 hours. ACS may be ST-elevation myocardial infarction (STEMI), non-STEMI (NSTEMI), or unstable angina (UA). Successful treatment with PCI is defined as achievement of <30% residual diameter stenosis of the target lesion assessed by visual inspection or quantitative coronary angiography and no in-hospital major adverse cardiac events (AMI or repeat coronary revascularisation of the target lesion). For ACS patients with ST-segment elevation, persistent ST-segment elevation of at least 0.1 mV in at least two contiguous leads or a new left bundle-branch block should be present. For ACS patients without ST-segment elevation, at least two of the following three criteria should be met: (i) ST-segment changes on electrocardiography, indicating ischemia; (ii) a positive test of a biomarker, indicating myocardial necrosis; or (iii) one of several risk factors (age ≥60 years; previous myocardial infarction or coronary artery bypass grafting; coronary artery disease with stenosis of ≥50% in at least two vessels; previous ischemic stroke, transient ischemic attack, carotid stenosis of at least 50%, or cerebral revascularization; diabetes mellitus; peripheral arterial disease; chronic renal dysfunction, defined as a creatinine clearance of <60 ml per minute per 1.73 m2 of body surface area).
* The patient must be able to give informed consent in accordance with ICH GCP guidelines and local legislation and/or regulations.

Exclusion Criteria:

* Mechanical or biological heart valve prosthesis;
* PCI with bare-metal stent insertion;
* Unsuccessful PCI (>30% residual stenosis of the target lesion);
* Cardiogenic shock during current hospitalization;
* Adverse bleeding or ischaemic event during current hospitalization;
* Anaemia (haemoglobin <10 g/dL) or thrombocytopenia (platelet count <100 x109/L) at screening,
* Severe renal impairment (creatinine clearance <30mL/min (estimated CrCl calculated by Cockcroft-Gault equation) at screening;
* Active liver disease at screening, as indicated by at least one of the following: persistent alanine aminotransferase (ALT) or aspartate transaminase (AST) >3-fold upper limit of normal (ULN), known active hepatitis C, known active hepatitis B, known active hepatitis A;
* Use of fibrinolytic agents within 24 hours of screening;
* Gastrointestinal bleeding within 1 month prior to screening unless, in the opinion of the Investigator, the cause has been permanently eliminated (e.g., by surgery);
* Major bleeding episode (reduction in the hemoglobin level of at least 2 g/dL, transfusion of at least two units of blood, or symptomatic bleeding in a critical area or organ), including life-threatening bleeding episode (symptomatic intracranial bleeding, bleeding with a decrease in the hemoglobin level of at least 5 g/dL or bleeding requiring transfusion of at least 4 units of blood or inotropic agents or necessitating surgery) within 1 month prior to screening;
* Stroke within 1 month prior to screening;
* Major surgery within 1 month prior to screening;
* Malignancy or radiation therapy within 6 months prior to screening unless, in the opinion of the Investigator, the estimated life expectancy is greater than 36 months;
* History of intraocular, spinal, retroperitoneal, or traumatic intra-articular bleeding unless the causative factor has been permanently eliminated or repaired;
* Hemorrhagic disorder or bleeding diathesis (e.g. von Willebrand disease, hemophilia A or B or other hereditary bleeding disorder, history of spontaneous intra-articular bleeding, history of prolonged bleeding after surgery/intervention);
* Past an organ transplant or patient on the waiting list for organ transplant;
* Need for continued treatment with systemic ketoconazole, itraconazole, posaconazole, cyclosporine, tacrolimus, dronedarone, rifampicin, phenytoin, carbamazepine, St. John's Wort or any cytotoxic/myelosuppressive therapy.
* Need for continued treatment with non-steroidal anti-inflammatory drugs (NSAIDs);
* Pre-menopausal women (last menstruation ≤1 year prior to screening) who: sre pregnant or breastfeeding or are not surgically sterile or are of childbearing potential and not practicing two acceptable methods of birth control, or do not plan to continue practicing an acceptable method of birth control throughout the trial. Acceptable methods of birth control are oral or parenteral (patch, injection, implant) hormonal contraception, which has been used continuously for at least one month prior to the first dose of study medication, intrauterine device or intrauterine system, double-barrier method of contraception (condom and occlusive cap or condom and spermicidal agent), male sterilization and complete sexual abstinence (if acceptable by local authorities). Periodic abstinence is not an acceptable method of contraception.
* Known allergy to dabigatran, ticagrelor, clopidogrel, aspirin, or to the excipients used for the tables of the drugs;
* Contraindications, in the Investigator's opinion to dabigatran, ticagrelor, clopidogrel, or aspirin;
* Participation in another trial with an investigational drug or device within the past 30 days preceding the screening visit (patients participating in an observational study only will not be excluded);
* Patients who are not willing or able to comply with the protocol requirements or considered unreliable by the Investigator concerning the requirements for follow-up during the study and/or compliance with study drug administration, who have a life expectancy less than the expected duration of the trial due to concomitant disease, or who have any condition which in the opinion of the Investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2230 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint - first major or clinically relevant non-major bleeding event, as defined by the ISTH | 24 months
  First major or clinically relevant non-major bleeding event, as defined by the International Society on Thrombosis and Haemostasis (ISTH)

SECONDARY OUTCOMES:
Secondary efficacy endpoint - thromboembolic events or death or unplanned revascularization; individual thromboembolic events; definite stent thrombosis | 24 months
  Composite efficacy endpoint of thromboembolic events (myocardial infarction, stroke, or systemic embolism) or death or unplanned revascularization (PCI or coronary artery bypass grafting); individual thromboembolic events (death, myocardial infarction, stroke, systemic embolism); definite stent thrombosis
Secondary safety endpoint - major bleeding events; clinically relevant non-major bleeding events; clinically relevant bleeding; minor and total bleeding; intracranial hemorrhage | 24 months
  major bleeding events (per ISTH); clinically relevant non-major bleeding events; clinically relevant bleeding (BARC ≥3 or TIMI major and minor); minor and total bleeding (ISTH, BARC, TIMI; total bleeding is the sum of all major and minor bleeds); intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Leszczyńska-Wiloch, PhD, Principal Investigator — Department of Non-Commercial Clinical Research, Medical University of Gdansk
Locations (1):
- Cardiac lntensive Care Unit, First Department of Cardiology, University Clinical Centre in Gdańsk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No